CLINICAL TRIAL: NCT01880684
Title: Validation of Capnography as a Predictor of Cardiac Output Change as Measured by FloTrac
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Andre Denault, MD FRCPC ABIM-CCM, Montreal Heart Institute
Other Study IDs: 13-1437
Record Dates: First submitted 2013-06-07; First posted 2013-06-19 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Hypovolemia; Cardiac Output, High; Cardiac Output, Low
Keywords: Thermodilution; Blood Volume; Cardiac Output; Leg; Capnography; Blood Pressure
MeSH Terms: conditions — Hypovolemia; Cardiac Output, High; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Passive Leg Rising

SUMMARY:
The aim of this study is to evaluate the correlation of capnography with non-invasive measurement of cardiac output with the FloTrac/EV1000 following a reversible fluid challenge, a passive leg raising maneuver, using thermodilution as the gold standard.

The main hypothesis is a correlation of 0.8 between the increasing of ETCO2 and the increasing of ejection volume measured by FloTrac/EV1000 following a passive leg raising maneuver.

DETAILED DESCRIPTION:
Data are collected on past medical illnesses, medication, type of surgery, abnormalities on pre-operative transesophageal echocardiogram and localisation of arterial line.

Before induction of anesthesia, an arterial line is installed. The agents of induction of anesthesia and doses are left to the discretion of the attending anesthesiologist. The trachea is intubated, anesthesia circuit and sidestream CO2 sensor were connected to the endotracheal tube and positive pressure ventilation begins with standardized parameters: control assisted mode with no inspiratory effort, tidal volume of 6-8 mL/kg, respiratory rate of 8-10/minute and PEEP of 5 mmHg. Modification of the ventilation parameters is not permitted before and during the PLR maneuvers. Isoflurane and propofol are used for the maintenance of anesthesia. A PA catheter (Paceport, Edwards Lifesciences, Irvine, California, USA) is inserted in the right internal jugular vein. If a femoral line is installed, the FloTrac/EV1000 is connected to the femoral line, if not, the radial line is used for mini-invasive continuous cardiac output monitoring. The a and v wave aspect and ratio of CVP waveform is noted. The RV waveform is inspected for signs of abnormalities such as a non-horizontal slope restrictive pattern (Figure xx)18. The transducers are all placed at the midthoracic level and a "flush test" is performed prior to CO measurements with the FloTrac/EV1000 to ensure absence of resonance or damping of the system.

At baseline, in the operating room before the first PLR maneuver, the heart rate, systolic, diastolic and mean arterial pressure, CVP value, CI measured in triplicate with the thermodilution method and the FloTrac derived variables are recorded. These variables include the CO indexed CO and SVV measured by the FloTrac/EV1000. The same variables are recorded at 1, 3 and 5 minutes after the beginning of PLR except CI by thermodilution which is measured again only once, at 3 minutes and EtCO2 which is recorded every 12 seconds. The EtCO2 curve is inspected at baseline and during the PLR maneuver to ensure the changes in EtCO2 were not related to changes in inspired CO2, ventilator or circuit malfunction or increase in airway resistance.

After weaning from CPB, the same measures are taken twice: with chest opened, when hemodynamic stability is achieved, and CPB canulas taken out and with chest closed.

In the ICU, two additional PLR maneuvers were executed with a 30 minutes interval in between. The set of measurements previously described are recorded. The use of an epicardial temporary pacemaker, vasopressors (doses and type), vasodilators (doses and type) are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more who have cardiac or aortic surgery

Exclusion Criteria:

* Pacemaker
* Lower limb amputation or absence of lower limb
* Moderate tricuspid insufficiency
* Preoperative arrythmia or prolonged arrythmia during data measurements
* Moderate aortic regurgitation
* Known deep vein thrombosis
* Intra-aortic balloon pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years old or more presenting for cardiac or aortic surgery at the Montreal Heart Institute.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Correlation between elevation in ETCO2 and cardiac output during a reversible fluid challenge, a passive leg raise | Participants will be followed from their arrival in the operating room until 2 hours post-operatively in the intensive care unit
  Correlation of 0.8 between the increase of ETCO2 and the increase of ejection volume measured by FloTrac/EV1000 following a passive leg raising maneuver

SECONDARY OUTCOMES:
Correlation between changes in indexed cardiac output measured by Flotrac/EV1000 and by thermodilution during a reversible fluid challenge, a passive leg raise | Participants will be followed from their arrival in the operating room until 2 hours post-operatively in the intensive care unit
Correlation between elevation in capnography and indexed cardiac output measured by thermodilution during a reversible fluid challenge, a passive leg raise | Participants will be followed from their arrival in the operating room until 2 hours post-operatively in the intensive care unit
Correlation between changes in capnography and indexed cardiac output measured by Flotrac/EV1000 during a reversible fluid challenge, a passive leg raise | Participants will be followed from their arrival in the operating room until 2 hours post-operatively in the intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] MARINO, Paul L. The ICU Book. Philadelphie, PA, Lippincott Williams & Wilkins, 2007, 1065 pages.
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Kumar A, Anel R, Bunnell E, Habet K, Zanotti S, Marshall S, Neumann A, Ali A, Cheang M, Kavinsky C, Parrillo JE. Pulmonary artery occlusion pressure and central venous pressure fail to predict ventricular filling volume, cardiac performance, or the response to volume infusion in normal subjects. Crit Care Med. 2004 Mar;32(3):691-9. doi: 10.1097/01.ccm.0000114996.68110.c9. PMID 15090949
- [Background] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Background] Tavernier B, Makhotine O, Lebuffe G, Dupont J, Scherpereel P. Systolic pressure variation as a guide to fluid therapy in patients with sepsis-induced hypotension. Anesthesiology. 1998 Dec;89(6):1313-21. doi: 10.1097/00000542-199812000-00007. PMID 9856704
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] Perel A. Assessing fluid responsiveness by the systolic pressure variation in mechanically ventilated patients. Systolic pressure variation as a guide to fluid therapy in patients with sepsis-induced hypotension. Anesthesiology. 1998 Dec;89(6):1309-10. doi: 10.1097/00000542-199812000-00005. No abstract available. PMID 9856702
- [Background] Lattik R, Couture P, Denault AY, Carrier M, Harel F, Taillefer J, Tardif JC. Mitral Doppler indices are superior to two-dimensional echocardiographic and hemodynamic variables in predicting responsiveness of cardiac output to a rapid intravenous infusion of colloid. Anesth Analg. 2002 May;94(5):1092-9, table of contents. doi: 10.1097/00000539-200205000-00007. PMID 11973168
- [Background] Tousignant CP, Walsh F, Mazer CD. The use of transesophageal echocardiography for preload assessment in critically ill patients. Anesth Analg. 2000 Feb;90(2):351-5. doi: 10.1097/00000539-200002000-00021. PMID 10648320
- [Background] Shibutani K, Muraoka M, Shirasaki S, Kubal K, Sanchala VT, Gupte P. Do changes in end-tidal PCO2 quantitatively reflect changes in cardiac output? Anesth Analg. 1994 Nov;79(5):829-33. doi: 10.1213/00000539-199411000-00002. PMID 7978395
- [Background] Isserles SA, Breen PH. Can changes in end-tidal PCO2 measure changes in cardiac output? Anesth Analg. 1991 Dec;73(6):808-14. doi: 10.1213/00000539-199112000-00023. PMID 1952183
- [Background] Maslow A, Stearns G, Bert A, Feng W, Price D, Schwartz C, MacKinnon S, Rotenberg F, Hopkins R, Cooper G, Singh A, Loring S. Monitoring end-tidal carbon dioxide during weaning from cardiopulmonary bypass in patients without significant lung disease. Anesth Analg. 2001 Feb;92(2):306-13. doi: 10.1097/00000539-200102000-00004. PMID 11159221
- [Background] Breukers RM, Sepehrkhouy S, Spiegelenberg SR, Groeneveld AB. Cardiac output measured by a new arterial pressure waveform analysis method without calibration compared with thermodilution after cardiac surgery. J Cardiothorac Vasc Anesth. 2007 Oct;21(5):632-5. doi: 10.1053/j.jvca.2007.01.001. Epub 2007 Apr 5. PMID 17905265
- [Background] Cannesson M, Musard H, Desebbe O, Boucau C, Simon R, Henaine R, Lehot JJ. The ability of stroke volume variations obtained with Vigileo/FloTrac system to monitor fluid responsiveness in mechanically ventilated patients. Anesth Analg. 2009 Feb;108(2):513-7. doi: 10.1213/ane.0b013e318192a36b. PMID 19151280
- [Background] Broch O, Renner J, Gruenewald M, Meybohm P, Schottler J, Steinfath M, Malbrain M, Bein B. A comparison of third-generation semi-invasive arterial waveform analysis with thermodilution in patients undergoing coronary surgery. ScientificWorldJournal. 2012;2012:451081. doi: 10.1100/2012/451081. Epub 2012 Jul 31. PMID 22919321
- [Background] Kusaka Y, Yoshitani K, Irie T, Inatomi Y, Shinzawa M, Ohnishi Y. Clinical comparison of an echocardiograph-derived versus pulse counter-derived cardiac output measurement in abdominal aortic aneurysm surgery. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):223-6. doi: 10.1053/j.jvca.2011.07.011. Epub 2011 Sep 15. PMID 21924632
- [Background] Su BC, Tsai YF, Cheng CW, Yu HP, Yang MW, Lee WC, Lin CC. Stroke volume variation derived by arterial pulse contour analysis is a good indicator for preload estimation during liver transplantation. Transplant Proc. 2012 Mar;44(2):429-32. doi: 10.1016/j.transproceed.2011.12.037. PMID 22410035
- [Background] Tsai YF, Su BC, Lin CC, Liu FC, Lee WC, Yu HP. Cardiac output derived from arterial pressure waveform analysis: validation of the third-generation software in patients undergoing orthotopic liver transplantation. Transplant Proc. 2012 Mar;44(2):433-7. doi: 10.1016/j.transproceed.2011.12.045. PMID 22410036
- [Background] McLean AS, Huang SJ, Kot M, Rajamani A, Hoyling L. Comparison of cardiac output measurements in critically ill patients: FloTrac/Vigileo vs transthoracic Doppler echocardiography. Anaesth Intensive Care. 2011 Jul;39(4):590-8. doi: 10.1177/0310057X1103900409. PMID 21823375
- [Background] Slagt C, de Leeuw MA, Beute J, Rijnsburger E, Hoeksema M, Mulder JW, Malagon I, Groeneveld AB. Cardiac output measured by uncalibrated arterial pressure waveform analysis by recently released software version 3.02 versus thermodilution in septic shock. J Clin Monit Comput. 2013 Apr;27(2):171-7. doi: 10.1007/s10877-012-9410-9. Epub 2012 Nov 15. PMID 23154918
- [Background] Biais M, Vidil L, Sarrabay P, Cottenceau V, Revel P, Sztark F. Changes in stroke volume induced by passive leg raising in spontaneously breathing patients: comparison between echocardiography and Vigileo/FloTrac device. Crit Care. 2009;13(6):R195. doi: 10.1186/cc8195. Epub 2009 Dec 7. PMID 19968880
- [Background] Mutoh T, Ishikawa T, Kobayashi S, Suzuki A, Yasui N. Performance of Third-generation FloTrac/Vigileo system during hyperdynamic therapy for delayed cerebral ischemia after subarachnoid hemorrhage. Surg Neurol Int. 2012;3:99. doi: 10.4103/2152-7806.100195. Epub 2012 Aug 27. PMID 23061015
- [Background] Rutlen DL, Wackers FJ, Zaret BL. Radionuclide assessment of peripheral intravascular capacity: a technique to measure intravascular volume changes in the capacitance circulation in man. Circulation. 1981 Jul;64(1):146-52. doi: 10.1161/01.cir.64.1.146. PMID 6786793
- [Background] Reich DL, Konstadt SN, Raissi S, Hubbard M, Thys DM. Trendelenburg position and passive leg raising do not significantly improve cardiopulmonary performance in the anesthetized patient with coronary artery disease. Crit Care Med. 1989 Apr;17(4):313-7. doi: 10.1097/00003246-198904000-00003. PMID 2702840
- [Background] THOMAS M, SHILLINGFORD J. THE CIRCULATORY RESPONSE TO A STANDARD POSTURAL CHANGE IN ISCHAEMIC HEART DISEASE. Br Heart J. 1965 Jan;27(1):17-27. doi: 10.1136/hrt.27.1.17. No abstract available. PMID 14242159
- [Background] Rocha P, Lemaigre D, Leroy M, Desfonds P, De Zuttere D, Liot F. Nitroglycerin-induced decrease of carbon monoxide diffusion capacity in acute myocardial infarction reversed by elevating legs. Crit Care Med. 1987 Feb;15(2):131-3. doi: 10.1097/00003246-198702000-00010. PMID 3100135
- [Background] Takagi S, Yokota M, Iwase M, Yoshida J, Hayashi H, Sotobata I, Koide M, Saito H. The important role of left ventricular relaxation and left atrial pressure in the left ventricular filling velocity profile. Am Heart J. 1989 Nov;118(5 Pt 1):954-62. doi: 10.1016/0002-8703(89)90230-5. PMID 2683699
- [Background] Gaffney FA, Bastian BC, Thal ER, Atkins JM, Blomqvist CG. Passive leg raising does not produce a significant or sustained autotransfusion effect. J Trauma. 1982 Mar;22(3):190-3. doi: 10.1097/00005373-198203000-00003. PMID 7069801
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Background] Preau S, Saulnier F, Dewavrin F, Durocher A, Chagnon JL. Passive leg raising is predictive of fluid responsiveness in spontaneously breathing patients with severe sepsis or acute pancreatitis. Crit Care Med. 2010 Mar;38(3):819-25. doi: 10.1097/CCM.0b013e3181c8fe7a. PMID 20016380
- [Background] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Background] Muller L, Toumi M, Bousquet PJ, Riu-Poulenc B, Louart G, Candela D, Zoric L, Suehs C, de La Coussaye JE, Molinari N, Lefrant JY; AzuRea Group. An increase in aortic blood flow after an infusion of 100 ml colloid over 1 minute can predict fluid responsiveness: the mini-fluid challenge study. Anesthesiology. 2011 Sep;115(3):541-7. doi: 10.1097/ALN.0b013e318229a500. PMID 21792056
- [Background] Monnet X, Bataille A, Magalhaes E, Barrois J, Le Corre M, Gosset C, Guerin L, Richard C, Teboul JL. End-tidal carbon dioxide is better than arterial pressure for predicting volume responsiveness by the passive leg raising test. Intensive Care Med. 2013 Jan;39(1):93-100. doi: 10.1007/s00134-012-2693-y. Epub 2012 Sep 19. PMID 22990869
- [Background] Denault AY, Haddad F, Jacobsohn E, Deschamps A. Perioperative right ventricular dysfunction. Curr Opin Anaesthesiol. 2013 Feb;26(1):71-81. doi: 10.1097/ACO.0b013e32835b8be2. PMID 23235519
- [Background] Madsen PL, Nielsen HB, Christiansen P. Well-being and cerebral oxygen saturation during acute heart failure in humans. Clin Physiol. 2000 Mar;20(2):158-64. doi: 10.1046/j.1365-2281.2000.00241.x. PMID 10735984
- [Background] Paquet C, Deschamps A, Denault AY, Couture P, Carrier M, Babin D, Levesque S, Piquette D, Lambert J, Tardif JC. Baseline regional cerebral oxygen saturation correlates with left ventricular systolic and diastolic function. J Cardiothorac Vasc Anesth. 2008 Dec;22(6):840-6. doi: 10.1053/j.jvca.2008.02.013. Epub 2008 May 12. PMID 18834789
- [Background] Sokol DK, Markand ON, Daly EC, Luerssen TG, Malkoff MD. Near infrared spectroscopy (NIRS) distinguishes seizure types. Seizure. 2000 Jul;9(5):323-7. doi: 10.1053/seiz.2000.0406. PMID 10933986
- [Background] Shojima M, Watanabe E, Mayanagi Y. Cerebral blood oxygenation after cerebrospinal fluid removal in hydrocephalus measured by near infrared spectroscopy. Surg Neurol. 2004 Oct;62(4):312-8; discussion 318. doi: 10.1016/j.surneu.2003.09.035. PMID 15451273
- [Background] Gracias VH, Guillamondegui OD, Stiefel MF, Wilensky EM, Bloom S, Gupta R, Pryor JP, Reilly PM, Leroux PD, Schwab CW. Cerebral cortical oxygenation: a pilot study. J Trauma. 2004 Mar;56(3):469-72; discussion 472-4. doi: 10.1097/01.ta.0000114274.95423.c0. PMID 15128115
- [Background] Vernieri F, Tibuzzi F, Pasqualetti P, Rosato N, Passarelli F, Rossini PM, Silvestrini M. Transcranial Doppler and near-infrared spectroscopy can evaluate the hemodynamic effect of carotid artery occlusion. Stroke. 2004 Jan;35(1):64-70. doi: 10.1161/01.STR.0000106486.26626.E2. Epub 2003 Dec 18. PMID 14684777
- [Background] Taillefer MC, Denault AY. Cerebral near-infrared spectroscopy in adult heart surgery: systematic review of its clinical efficacy. Can J Anaesth. 2005 Jan;52(1):79-87. doi: 10.1007/BF03018586. PMID 15625262
- [Background] Nagdyman N, Ewert P, Peters B, Miera O, Fleck T, Berger F. Comparison of different near-infrared spectroscopic cerebral oxygenation indices with central venous and jugular venous oxygenation saturation in children. Paediatr Anaesth. 2008 Feb;18(2):160-6. doi: 10.1111/j.1460-9592.2007.02365.x. PMID 18184248
- [Background] Boulain T, Achard JM, Teboul JL, Richard C, Perrotin D, Ginies G. Changes in BP induced by passive leg raising predict response to fluid loading in critically ill patients. Chest. 2002 Apr;121(4):1245-52. doi: 10.1378/chest.121.4.1245. PMID 11948060
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454